CLINICAL TRIAL: NCT00748215
Title: Phase II, Randomized, Double Blind Comparison of CASAD vs. Placebo for the Treatment and Prevention of Diarrhea in Patients With Metastatic Colorectal Cancer
Brief Title: Calcium Aluminosilicate Anti-Diarrheal in Treating and Preventing Diarrhea in Patients With Metastatic Colorectal Cancer Receiving Irinotecan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MDA-2008-0005; MDA-2008-0005; CDR0000612205 (Other: NCI Clinical Trials)
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Chemotherapeutic Agent Toxicity; Colorectal Cancer; Diarrhea
Keywords: diarrhea; chemotherapeutic agent toxicity; recurrent colon cancer; recurrent rectal cancer; stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Diarrhea; Colonic Neoplasms; Rectal Neoplasms | interventions — Calcium Aluminosilicate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: CASAD (Experimental): Oral calcium aluminosilicate anti-diarrheal (CASAD) 4 times daily for 6 weeks in the absence of disease progression or unacceptable toxicity. Participants who develop grade 3 or 4 diarrhea may receive CASAD for an additional 6 weeks.
  Interventions: Drug: calcium aluminosilicate anti-diarrheal
- Arm II: Placebo (Placebo Comparator): Oral placebo 4 times daily for 6 weeks in the absence of disease progression or unacceptable toxicity. Participants who develop grade 3 or 4 diarrhea may then receive CASAD for 6 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: calcium aluminosilicate anti-diarrheal — Given orally
  Arms: Arm I: CASAD
Other: placebo — Given orally
  Arms: Arm II: Placebo

SUMMARY:
RATIONALE: Calcium aluminosilicate anti-diarrheal (CASAD) may help treat and prevent diarrhea caused by irinotecan. It is not yet known whether CASAD is more effective than a placebo in treating and preventing diarrhea in patients receiving irinotecan.

PURPOSE: This randomized phase II trial is studying CASAD to see how well it works compared with a placebo in treating and preventing diarrhea in patients with metastatic colorectal cancer receiving irinotecan.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the efficacy of calcium aluminosilicate anti-diarrheal (CASAD) versus placebo in reducing the incidence of grade 3 or 4 diarrhea in patients with metastatic colorectal cancer receiving an irinotecan-based chemotherapy regimen.

Secondary

* To compare stools per day in patients treated with these drugs.
* To compare chemotherapy dose reductions and delays due to diarrhea in patients treated with these drugs.
* To compare quality of life of patients treated with these drugs.
* To compare the safety of these drugs in these patients.
* To compare the incidence of grade 3 or 4 diarrhea in patients treated with these drugs.

OUTLINE: This is a multicenter study. Patients are stratified according to chemotherapy regimen (irinotecan hydrochloride in combination with fluorouracil and/or biologic therapy vs irinotecan hydrochloride alone). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral calcium aluminosilicate anti-diarrheal (CASAD) 4 times daily for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients who develop grade 3 or 4 diarrhea and are removed from the study may receive CASAD for an additional 6 weeks.
* Arm II: Patients receive oral placebo 4 times daily for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients who develop grade 3 or 4 diarrhea and are removed from the study may then receive CASAD for 6 weeks.

Patients undergo quality-of-life assessment at baseline and at weeks 3, 5, and 6.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal cancer

  * Metastatic disease
* Scheduled to receive irinotecan hydrochloride alone or in combination with fluorouracil, cetuximab, leucovorin calcium, or other biological therapy (including bevacizumab)
* No uncontrolled brain metastasis

  * Previously treated brain metastasis allowed

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) > 1,000/mm³
* Platelet count > 100,000/mm³
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST or SGOT) and/or alanine aminotransferase (ALT or SGPT) < 2.5 times ULN (< 5 times ULN if liver metastasis is present)
* Alkaline phosphatase < 2.5 times ULN
* Creatinine clearance > 35 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known UDP-glucuronosyltransferase 1A1 (UGT1A1) deficiency with homozygotes.
* No known history of Gilbert's disease
* No diarrhea > grade 1
* No serious illness or medical condition, including any of the following:

  * Uncontrolled congestive heart failure
  * Uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg)
  * Uncontrolled arrhythmia
  * Active angina pectoris
  * Symptomatic heart disease according to New York Heart Association(NYHA) class II-IV
* No serious uncontrolled active infection
* No existing colostomy or ileostomy
* Not able to take and document oral study medications
* No history of allergies to irinotecan hydrochloride
* No history of significant neurological or psychiatric disorders that would preclude giving consent or participating in study treatment or follow up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior treatment for metastatic disease allowed
* At least 4 weeks since prior irinotecan
* More than 2 weeks since prior chemotherapy

  * Irinotecan alone or in combination with other chemotherapy or biologic agents allowed
* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy
* No concurrent medication schedule that does not permit a 2-hour window between administration of calcium aluminosilicate anti-diarrheal (CASAD) and other medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-02-04 (Actual); Primary Completion 2014-08-12 (Actual); Study Completion 2014-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian K. Kee, MD, Study Chair — M.D. Anderson Cancer Center; Michael J. Fisch, MD, MPH, FACP, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- See also: Related Info — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 04, 2009 to May 3, 2012. All recruitment done at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the original 100 patients enrolled and randomized to the 6 week intervention period, 39 patients would go on to take open label CASAD; 22 patients from the CASAD arm and 17 patients from the placebo arm. These patients were added as a Milestone on the Participant Flow sheet. 8 patients received open label for <21 days; 31 patients received open label CASAD for >21 days.
Groups:
- Arm I: Calcium Aluminosilicate Anti-Diarrheal (CASAD): Oral calcium aluminosilicate anti-diarrheal (CASAD) 4 times daily for 6 weeks in the absence of disease progression or unacceptable toxicity. Participants who develop grade 3 or 4 diarrhea may receive CASAD for an additional 6 weeks.
Period: Overall Study
Arm/Group | Arm I: Calcium Aluminosilicate Anti-Diarrheal (CASAD) | Arm II: Placebo
Started | 50 | 50
Open Label CASAD After Initial 6 Weeks Intervention | 22 | 17
Completed | 41 | 32
Not Completed | 9 | 18
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Treatment change | 2 | 1
Not completed — Change in patient condition | 0 | 3
Not completed — Non-compliant | 0 | 2
Not completed — Adverse Event | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Calcium Aluminosilicate Anti-Diarrheal (CASAD) | Arm II: Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Full Range); unit: Years] | 57 [20 to 83] | 56 [26 to 81] | 56.5 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 29 | 25 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 45 | 44 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 42 | 41 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Baseline Bowel Assessment (BBA) [Count of Participants; unit: Participants] — The number of normal bowel movements/stools in a day.
  Participants
    < 1 Per Day | 7 | 6 | 13
    < 1 -3 Per Day | 7 | 3 | 10
    < >3 Per Day | 27 | 34 | 61
    Other | 3 | 3 | 6
Baseline Ostomy Bowel Assessment (BOBA) [Count of Participants; unit: Participants] — The number of times in a 24-hour day change the ostomy bag
  Participants
    2-3 times | 3 | 3 | 6
    4-6 times | 2 | 0 | 2
    >6 times | 0 | 0 | 0
    Other | 2 | 1 | 3
Baseline Bowel Assessment (BBA) [Count of Participants; unit: Participants] — Number of participants with recent alternating constipation/diarrhea or recent changes in bowel pattern
  Participants
    No | 7 | 6 | 13
    Yes, some | 24 | 32 | 56
    Yes, significant | 11 | 8 | 19
    Not answered | 2 | 0 | 2
Baseline Bowel Assessment (BBA) [Count of Participants; unit: Participants] — Form of bowel movements/stools
  Participants
    Hard difficult to pass | 8 | 9 | 17
    Well-formed, easy to pass | 4 | 2 | 6
    Loose | 25 | 29 | 54
    Very loose and watery | 7 | 6 | 13
    Not answered | 0 | 3 | 3
Baseline Bowel Assessment (BBA) [Count of Participants; unit: Participants] — How often is the ostomy bag is changed
  Participants
    1/4 Full | 0 | 1 | 1
    1/3 Full (recommended) | 4 | 1 | 5
    1/2 Full | 1 | 1 | 2
    Other | 1 | 0 | 1
Baseline Ostomy Bowel Assessment (BOBA) [Count of Participants; unit: Participants] — Do you normally measure the amount of your ostomy output? If so, what do you consider your normal volume of output in a 24-hour day?
  Participants
    Does not measure output | 6 | 4 | 10
    <200 ml/day | 0 | 0 | 0
    200-600 ml/day (typical) | 0 | 0 | 0
    600-1000 ml/day | 0 | 0 | 0
    >1000 ml/day | 0 | 0 | 0
Baseline Ostomy Bowel Assessment (BOBA) [Count of Participants; unit: Participants] — Have the participant had any recent alternating constipation/diarrhea or recent changes in bowel pattern?
  Participants
    No | 4 | 4 | 8
    Yes, some | 1 | 0 | 1
    Yes, significant | 1 | 0 | 1
Baseline Ostomy Bowel Assessment (BOBA) [Count of Participants; unit: Participants] — On average, how well-formed are your bowel movements/stool?
  Participants
    Well-formed, easy to pass | 0 | 0 | 0
    Semi-formed (peanut butter consistency) | 1 | 3 | 4
    Loose (pudding, cake batter consistency) | 2 | 1 | 3
    Very loose and watery | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3/4 Diarrhea
Description: One hundred patients were randomized equally between CASAD and placebo arms in order to assess whether CASAD was efficacious in preventing grade 3/4 diarrhea within 6 weeks for each arm compared. Bayesian futility monitoring in the study with a recommendation to stop the trial for futility if it became clear that CASAD was not better than placebo.
Time Frame: First 6 weeks from baseline in initial intervention with CASAD or PLACEBO
Population: Patients who experienced any diarrhea during the intervention period and patients who experienced Grade 3/4 diarrhea during the intervention period.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Calcium Aluminosilicate Anti-Diarrheal (CASAD) | Arm II: Placebo
Number analyzed (Participants) | 49 | 46
Participants
  Any diarrhea in first 6 weeks | 27 | 26
  Grade 3/4 diarrhea in first 6 weeks | 7 | 3

ADVERSE EVENTS:
Time Frame: Baseline at enrollment through 30 days following being taken off treatment for each participant, an average of 10 weeks
Description: An adverse event (AE) is any condition that appears or worsens after the subject is enrolled in an investigational study. AEs will be graded by numerical score according to the NCI Common Terminology Criteria Adverse Events (CTCAE)
Arm/Group | Arm I: Calcium Aluminosilicate Anti-Diarrheal (CASAD) | Arm II: Placebo
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 4/50 | 9/50
Other Adverse Events (participants affected / at risk) | 50/50 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Calcium Aluminosilicate Anti-Diarrheal (CASAD) (N=50) | Arm II: Placebo (N=50)
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Obstruction (Gastrointestinal disorders) | 0 | 2
Febrile Neutropenia (Infections and infestations) | 1 | 1
Abdominal Pain (General disorders) | 0 | 2
Renal Failure (Renal and urinary disorders) | 0 | 1
Fracture - skull (Musculoskeletal and connective tissue disorders) | 0 | 1
Hemorrhage - intracranial (Nervous system disorders) | 0 | 1
Creatinine - elevated (Renal and urinary disorders) | 0 | 1
Abdominal Distention (Gastrointestinal disorders) | 0 | 1
Dehydration (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Calcium Aluminosilicate Anti-Diarrheal (CASAD) (N=50) | Arm II: Placebo (N=50)
Abdominal distention (Gastrointestinal disorders) | 2 | 2
Abdominal pain (General disorders) | 7 | 9
Act prtl thromboplast t prolonged (Blood and lymphatic system disorders) | 0 | 2
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Agitation (Nervous system disorders) | 2 | 0
Alanine Aminotransferase increase (Metabolism and nutrition disorders) | 3 | 3
Alkaline phosphatase increase (Metabolism and nutrition disorders) | 5 | 6
Allergic reaction (Immune system disorders) | 1 | 0
Allergic rhinitis (Immune system disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 7
Anal pain (General disorders) | 1 | 0
Anemia (Metabolism and nutrition disorders) | 10 | 12
Anorexia (Gastrointestinal disorders) | 14 | 6
Anxiety (Nervous system disorders) | 4 | 6
Arthralgia (Immune system disorders) | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspartate aminotransferase increase (Metabolism and nutrition disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Back pain (General disorders) | 4 | 1
Bloating (Gastrointestinal disorders) | 2 | 1
Blood bilirubin increase (Metabolism and nutrition disorders) | 2 | 3
Bone pain (General disorders) | 0 | 1
Bruising (Skin and subcutaneous tissue disorders) | 0 | 1
Buttock pain (General disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Confusion (Nervous system disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 23 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Creatinine increase (Metabolism and nutrition disorders) | 1 | 5
Dehydration (Gastrointestinal disorders) | 7 | 3
Depr level of consciousness (Nervous system disorders) | 0 | 1
Depression (Nervous system disorders) | 7 | 5
Diarrhea (Gastrointestinal disorders) | 31 | 0
Dizziness (Nervous system disorders) | 6 | 3
Dry mouth (Gastrointestinal disorders) | 7 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Dysgeusia (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 0
Edema limbs (Cardiac disorders) | 3 | 4
Endocrine disorders (Endocrine disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Eye disorders (Eye disorders) | 1 | 2
Eyelid function disorder (Eye disorders) | 1 | 0
Fatigue (General disorders) | 29 | 21
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Fever (General disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 5 | 4
Flushing (Immune system disorders) | 2 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastroesophageal reflux (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 9 | 7
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 1
Gen disorders & admin site condition (General disorders) | 5 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Genital edema (Reproductive system and breast disorders) | 1 | 0
Glucose intolerance (Endocrine disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 0
Hematuria (Reproductive system and breast disorders) | 1 | 1
Hemoglobin increased (Metabolism and nutrition disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 4 | 1
Hiccups (Gastrointestinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hot flashes (Reproductive system and breast disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 3 | 7
Hypomagnesmia (Metabolism and nutrition disorders) | 1 | 5
Hyponatremia (Metabolism and nutrition disorders) | 5 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypothryoidism (Endocrine disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
INR increase (Metabolism and nutrition disorders) | 1 | 0
Immune system disorders (Immune system disorders) | 2 | 0
Infections and infestations (Infections and infestations) | 4 | 3
Insomnia (Nervous system disorders) | 4 | 5
Intestinal stoma obstruction (Gastrointestinal disorders) | 0 | 1
Investigations (Investigations) | 1 | 4
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Lymphocyte count decrease (Metabolism and nutrition disorders) | 5 | 2
Malaise (General disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 1
Metabolism & nurtition disorders (Metabolism and nutrition disorders) | 3 | 1
Mucosal infection (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 8 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 23 | 25
Neck pain (General disorders) | 2 | 0
Nervous system disorders (Nervous system disorders) | 6 | 3
Neutrophil count decrease (Metabolism and nutrition disorders) | 6 | 8
Obesity (Gastrointestinal disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 2
Oral dysethesia (Gastrointestinal disorders) | 0 | 1
Oral pain (General disorders) | 0 | 2
Pain (General disorders) | 11 | 9
Pain in extremity (General disorders) | 2 | 3
Palmar-plantar erythrodysesthias (Skin and subcutaneous tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 3 | 1
Paronychia (Infections and infestations) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Peripheral sensory neruopathy (Nervous system disorders) | 11 | 4
Platelet count descreased (Metabolism and nutrition disorders) | 3 | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 2
Renal and urinary disorders (Reproductive system and breast disorders) | 1 | 2
Respiratory, thoracic & mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Reproductive system & breast disorders (Reproductive system and breast disorders) | 0 | 1
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 8 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Somnolence (Nervous system disorders) | 2 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stomach pain (General disorders) | 2 | 0
Thromboembolic event (Blood and lymphatic system disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Urinary incontinence (Reproductive system and breast disorders) | 0 | 1
Urinary retention (Reproductive system and breast disorders) | 1 | 0
Urinary tract infection (Reproductive system and breast disorders) | 1 | 1
Vascular disorders (Cardiac disorders) | 1 | 3
Vaginal dryness (Reproductive system and breast disorders) | 0 | 1
Voice changes (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 13 | 16
Watering eyes (Immune system disorders) | 1 | 0
Weight gain (Investigations) | 0 | 1
Weight loss (Investigations) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wound complication (Skin and subcutaneous tissue disorders) | 0 | 1
White blood cell decreased (Metabolism and nutrition disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes